CLINICAL TRIAL: NCT00388206
Title: An Observational Study of Avastin (Bevacizumab) in Combination With Chemotherapy for Treatment of Metastatic or Locally Advanced and Unresectable Colorectal Cancer and Locally Advanced or Metastatic Non-Small Cell Lung Cancer (Excluding Predominant Squamous Cell Histology)
Brief Title: A Study of Avastin in Combination With Chemotherapy for Treatment of Colorectal Cancer and Non-Small Cell Lung Cancer (ARIES)
Acronym: ARIES
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AVF3991n
Record Dates: First submitted 2006-10-12; First posted 2006-10-16 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer; Non-Small Cell Lung Cancer
Keywords: NSCLC; Avastin; anti-VEGF; lung cancer; colorectal cancer; ARIES; Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and tumor

SUMMARY:
This is an observational study designed to follow patients with metastatic or locally advanced and unresectable CRC or locally advanced or metastatic NSCLC (excluding predominant squamous histology) who are receiving Avastin in combination with first-line chemotherapy. Second-line metastatic CRC patients are also eligible. Patients who started their Avastin containing therapy <4 months prior to enrollment are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Metastatic or locally advanced and unresectable CRC or locally advanced or metastatic NSCLC (excluding predominant squamous histology)
* Eligible for Avastin as a component of intended therapy
* First-line chemotherapy (or second-line chemotherapy for CRC) plus Avastin initiated ≤ 4 months prior to study enrollment

Exclusion Criteria:

* Any medical condition, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a patient's ability to provide informed consent or comply with the treatment and follow-up, as specified by the investigator
* Enrollment in a blinded, placebo-controlled bevacizumab trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 3998 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Wozniak AJ, Kosty MP, Jahanzeb M, Brahmer JR, Spigel DR, Leon L, Fish S, Flick ED, Hazard SJ, Lynch TJ Jr. Clinical outcomes in elderly patients with advanced non-small cell lung cancer: results from ARIES, a bevacizumab observational cohort study. Clin Oncol (R Coll Radiol). 2015 Apr;27(4):187-96. doi: 10.1016/j.clon.2014.12.002. Epub 2015 Jan 7. PMID 25576353
- [Derived] Douillard JY, Ostoros G, Cobo M, Ciuleanu T, Cole R, McWalter G, Walker J, Dearden S, Webster A, Milenkova T, McCormack R. Gefitinib treatment in EGFR mutated caucasian NSCLC: circulating-free tumor DNA as a surrogate for determination of EGFR status. J Thorac Oncol. 2014 Sep;9(9):1345-53. doi: 10.1097/JTO.0000000000000263. PMID 25122430
- [Derived] Lynch TJ Jr, Spigel DR, Brahmer J, Fischbach N, Garst J, Jahanzeb M, Kumar P, Vidaver RM, Wozniak AJ, Fish S, Flick ED, Leon L, Hazard SJ, Kosty MP; ARIES Study Investigators. Safety and effectiveness of bevacizumab-containing treatment for non-small-cell lung cancer: final results of the ARIES observational cohort study. J Thorac Oncol. 2014 Sep;9(9):1332-9. doi: 10.1097/JTO.0000000000000257. PMID 25122429